CLINICAL TRIAL: NCT05272228
Title: The Single-centre, Randomized, Comparative Single-dose Bioavailability Clinical Study of Different Coenzyme Q10 Products
Brief Title: Comparative Single-dose Bioavailability Clinical Study of Different Coenzyme Q10 Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Biovis d.o.o. (Unknown)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Associate Professor, PhD, University of Primorska
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: CoenzymeQ10
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Coenzyme Q Deficiency
Keywords: coenzyme Q10; single dose bioavailability
MeSH Terms: conditions — Coenzyme Q10 Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coenzyme Q10 (ubiquinone) (Active Comparator): Synonyms: Co-Q10; Ubiquinone; Ubidecarenone; 2,5-Cyclohexadiene-1,4-dione, 2- [(2E,6E,10E,14E,18E,22E,26E,30E,34E)-3,7,11,15,19,23,27,31,35,39-decamethyl-,6,10,14,18,22,26,30,34,38- tetracontadecaenyl]-5,6-dimethoxy-3-methyl CAS number: 303-98-0 Molecular formula: C59H90O4 USP standard Content: Co-Q10 (ubiquinone), bulking agent (maltodextrin), capsule (HPCM- hydroxypropyl methyl cellulose), anti-adherents (magnesium stearate and anhydrous silica) Dosage: 2 capsules, total 100 mg Co-Q10
  Interventions: Dietary Supplement: Dietary supplement - standard product
- Q10 MICROENCAPSULATED (Experimental): IP1:Q10 MICROENCAPSULATED. ENG: Ingredient BMT® Coenzyme Q10 Content Co-Q10 (ubiquinone), stabiliser (gum arabic), bulking agent (maltodextrin), capsule (HPCM- hydroxypropyl methyl cellulose), olive oil, corn starch, anti-adherents (magnesium stearate and anhydrous silica), acidity regulator (citric acid, acetic acid) HPMC capsules, size '0', 50 mg/capsule Dosage: 2 capsule, total 100 mg Co-Q10
  Interventions: Dietary Supplement: Dietary supplement - Investigational product IP1
- Final formulated product BQSM® (Experimental): IP2: Final formulated product BQSM® Ingredients: Rosehip (Rosa canina) fruit extract standardised to min. 70 % of vitamin C (L-ascorbic acid), capsule (HPCM- hydroxypropyl methyl cellulose), BMT® Coenzyme Q10 (ubiquinone), vitamin E (D-alfa tocopheryl acetate), vitamin A (retinyl acetate), L-selenomethionine, bulking agent (maltodextrin), stabiliser (gum arabic), olive oil, corn starch, anti-adherents (magnesium stearate and anhydrous silica), acidity regulator (citric acid, acetic acid) HPMC capsule, size '0', 50 mg/capsule Dosage: 2 capsule, total 100 mg Co-Q10
  Interventions: Dietary Supplement: Dietary supplement - Investigational product IP2

INTERVENTIONS:
Dietary Supplement: Dietary supplement - standard product — Single dose intervention with Standard product Coenzyme Q10 (ubiquinone) 2 capsules - 100 mg total coenzyme Q10
  Arms: Coenzyme Q10 (ubiquinone)
Dietary Supplement: Dietary supplement - Investigational product IP1 — Single dose intervention with Investigational product IP1; Q10 MICROENCAPSULATED 2 capsules - 100 mg total coenzyme Q10
  Arms: Q10 MICROENCAPSULATED
Dietary Supplement: Dietary supplement - Investigational product IP2 — Single dose intervention with Investigational product IP2; Final formulated product BQSM® 2 capsules - 100 mg total coenzyme Q10
  Arms: Final formulated product BQSM®

SUMMARY:
The randomized, open-label, three period crossover single-dose bioavailability study with three coenzyme Q10 products

DETAILED DESCRIPTION:
The randomized, open-label, three period crossover single-dose bioavailability study with three coenzyme Q10 products will include 25 subjects who will test three different coenzyme Q10 products. Serum concentration of coenzyme Q10 will be measured.

ELIGIBILITY:
Inclusion Criteria:

* subject informed consent form
* aged between 40 and 55 years old
* body mass for women 65± 5 kg and for men 85± 5 kg
* non-smoking
* healthy, without cardio-vascular diseases, diabetes, neurodegenerative diseases
* absence of any prescribed medication during the study
* willing to avoid a consumption of any food supplements at least 2 weeks before and during the study
* willing to study all study procedures

Exclusion Criteria:

* cardio-vascular diseases,
* diabetes,
* neurodegenerative diseases,
* gastrointestinal disorders
* hypotension
* pregnancy
* breast-feeding
* intake of any prescribed medication within two week of the beginning of the study
* intake of any food supplements within two week of the beginning of the study
* drug or alcohol abuse

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Serum coenzyme Q10 concentrations | 0,2,4,6,8,12 and 24 hours after ingestion
  Serum coenzyme Q10 concentrations will me measured in all three different coenzyme Q10 products with ELISA kit for coenzyme Q10

CONTACTS AND LOCATIONS:
Overall Officials: Zala Jenko-Pražnikar, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University of Primorska, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No